CLINICAL TRIAL: NCT05059548
Title: Sex Difference Effects on Postoperative Sleep, Inflammation and Cognition in Patients Undergoing General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, principal investigator, Shengjing Hospital
Other Study IDs: Sex, cognition, inflammation
Record Dates: First submitted 2021-09-12; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Sex Differences; Postoperative Sleep Quality; Postoperative Pain; Inflammation Function; Postoperative Cognitive Function
MeSH Terms: conditions — Pain, Postoperative | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male Group: Video-Assisted Thoracoscopic Surgery patients receive Video-Assisted Thoracoscopic Surgery under general anesthesia
  Interventions: Other: Video-Assisted Thoracoscopic Surgery
- Female Group: Video-Assisted Thoracoscopic Surgery patients receive Video-Assisted Thoracoscopic Surgery under general anesthesia
  Interventions: Other: Video-Assisted Thoracoscopic Surgery

INTERVENTIONS:
Other: Video-Assisted Thoracoscopic Surgery — patients receive Video-Assisted Thoracoscopic Surgery under general anesthesia

SUMMARY:
Video-Assisted Thoracoscopic Surgery(VATS) is among the most common and disabling persistent pain and inflammation conditions, with increasing prevalence in the developed world, and affects women to a greater degree than men. And sleep disruption also remains a challenging problem in surgical settings. Postoperative sleep disturbances (POSD) are defined as changes in the sleep structure and quality of patients during the early stages after surgery, which are manifested as significantly shortened rapid eye movement (REM) sleep, prolonged awake time, and sleep fragmentation. Long-term POSD may increase the risk of postoperative delirium or cognitive dysfunction and delay recovery, thereby worsening the patient's physical condition. The aim of the study was to investigate the effect of sex differences on postoperative pain, inflammation, sleep quality and cognitive function among patients who have undergone video-assisted thoracoscopic surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* ASA I-III
* under general anesthesia

Exclusion Criteria:

* patients with central nervous system and mental diseases;
* patients with preoperative sleep disturbances;
* patients with a history of sedative, analgesic, or antidepression drug use;
* patients with sleep apnea or moderate and severe obstructive sleep apneahypopnea syndrome;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing video-assisted thoracoscopic surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
sleep quality of one night before surgery | one night before surgery
  use the athens insomnia scale to evaluate subjective sleep quality (0 to 24 points, with ≥ 6 points indicating a diagnosis of insomnia)
sleep quality of first night after surgery | first night after surgery
  use the athens insomnia scale to evaluate subjective sleep quality (0 to 24 points, with ≥ 6 points indicating a diagnosis of insomnia)
sleep quality of third night after surgery | third night after surgery
  use the athens insomnia scale to evaluate subjective sleep quality (0 to 24 points, with ≥ 6 points indicating a diagnosis of insomnia)
preoperative inflammation function | three days before surgery
  evaluate systemic immune inflammation index (SII) before operation
preoperative inflammation function | three days before surgery
  evaluate neutrophil / lymphocyte ratio (NLR)before operation
preoperative inflammation function | three days before surgery
  evaluate platelet / lymphocyte ratio (PLR) before operation
preoperative inflammation function | three days before surgery
  evaluate monocyte / lymphocyte ratio (MLR) before operation
postoperative inflammation function | three days after surgery
  evaluate systemic immune inflammation index (SII) after operation
postoperative inflammation function | three days after surgery
  evaluate neutrophil / lymphocyte ratio (NLR) after operation
postoperative inflammation function | three days after surgery
  evaluate platelet / lymphocyte ratio (PLR) after operation
postoperative inflammation function | three days after surgery
  evaluate monocyte / lymphocyte ratio (MLR) after operation
neuropsychological test | Neuropsychological tests were carried out the day before and 5 to 7 days after surgery. The second neuropsychological test time for control subjects was 6 to 9 d
  The neuropsychological test battery included the tests used to evaluate patients for delayed neurocognitive recovery in the International Study of Post-Operative Cognitive Dysfunction: (1) word learning: visual verbal learning test based on the Rey's auditory recall of words; (2) word recall: the number or words recalled from visual verbal learning trials after a 20-min delay; (3) cognitive flexibility: including trail making test A and B; (4) distractibility: Stroop color word interference test; and (5) working memory: letter-digit coding. If a patient exhibited delirium at a testing time, neuropsychological evaluation was postponed 3 days.

SECONDARY OUTCOMES:
visual analog scale(VAS) score after surgery | 24 hours after surgery
  evaluate VAS (0-10 points)score 24 hours after surgery
postoperative adverse effects | 24 hours after surgery
  evaluate postoperative adverse effect 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: junchao zhu, Study Director — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China